CLINICAL TRIAL: NCT06339710
Title: Double Blind, Phase III Randomized,Safety and Efficacy Non-inferiority Trial to Evaluate Two Short Benznidazole Regimens for the Treatment of Adults in the Chronic Phase of Chagas Disease in Its Indeterminate and Mild Cardiac Forms in Bolivia and Colombia
Brief Title: Short Benznidazole Regimen for Chronic Phase Chagas Disease Patients
Acronym: Benlatino
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was finalized due to major administrative and contractual delays.
Sponsor: Evandro Chagas Institute of Clinical Research (Other)
Collaborators: Andrea Silvestre de Sousa (Unknown)
Responsible Party: Principal Investigator, Israel Molina, Principal Investigator, Evandro Chagas Institute of Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1288-5508
Record Dates: First submitted 2024-02-15; First posted 2024-04-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Chagas Disease
Keywords: Chagas disease; Short treatment; Benznidazole
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short treatment 1 (Experimental): benznidazole 300 mg daily for the first 2 weeks plus placebo for the last 6 weeks or
  Interventions: Drug: benznidazole 300 mg daily 8 weeks
- Short Treatment 2 (Experimental): benznidazole 300 mg daily for the first 4 weeks plus placebo for the last 4 weeks
  Interventions: Drug: benznidazole 300 mg daily 8 weeks
- Standard treatment (Active Comparator): benznidazole 300 mg daily for 8 weeks
  Interventions: Drug: benznidazole 300 mg daily 8 weeks

INTERVENTIONS:
Drug: benznidazole 300 mg daily 8 weeks — 672 participants will be randomly assigned to receive the standard-dose of benznidazole (300 mg daily for 8 weeks) or the short experimental regimens (benznidazole 300 mg daily for the first 2 weeks plus placebo for the last 6 weeks or benznidazole 300 mg daily for the first 4 weeks plus placebo for the last 4 weeks)
  Other Names: benznidazole 300 mg daily for the first 2 weeks plus placebo for the last 6 weeks; benznidazole 300 mg daily for the first 4 weeks plus placebo for the last 4 weeks

SUMMARY:
Multicentric study on Chagas disease that seeks to evaluate a new treatment regimen using the drug benznidazole. Currently, existing treatment regimens are long and have frequent side effects, which leads to a high dropout rate among patients. The research proposes testing two shorter benznidazole regimens to see if they are as effective as standard treatment, but with fewer side effects.

The study will have 672 participants and will be carried out in four locations, Bolivia and Colombia. The objective is to analyze the efficacy and safety of new treatment regimens, evaluating the parasitological response in comparison with standard treatment. In addition, an economic assessment will be carried out to analyze direct and indirect costs, including procedures associated with the management of adverse events.

DETAILED DESCRIPTION:
Chagas disease is a major cause of heart disease, morbidity, and premature loss of life in the Americas. Eliminating the Trypanosoma cruzi parasite using antitrypanosomal drugs has shown to produce cure in children, halt future congenital transmission, and reduce morbidity from the disease. However, the current treatment regimens are lengthy (60 days) and entail frequent side effects, causing about 20% of patients to drop out of treatment, and discouraging others from starting. Recent research found that a reduced treatment of benznidazole still has adequate efficacy with few side effects.

In this international, multicenter, double-blind, phase III, placebo-controlled study, 672 participants will be randomly assigned to receive the standard-dose of benznidazole (300 mg daily for 8 weeks) or the short experimental regimens (benznidazole 300 mg daily for the first 2 weeks plus placebo for the last 6 weeks or benznidazole 300 mg daily for the first 4 weeks plus placebo for the last 4 weeks). Efficacy will be assessed considering a non-inferiority design and through the detection of parasite deoxyribonucleic acid (DNA) through molecular biology (Polymerase Chain Reaction - PCR). Meanwhile, safety will be evaluated through a superiority design, with the aim to find the new regimen as effective as the standard one, but superior in terms of safety. An intention-to-treat analysis will be performed, and statistical significance will be set at 0.025 for the non-inferiority outcome (positive PCR) and 0.05 for the superiority outcome.

The study population will be adult participants, 18 years or older, with chronic Chagas disease in its indeterminate or mild cardiac forms, with a positive diagnosis from two serological assays. The trial will be conducted in four sites: two in Bolivia, and two in Colombia. The primary endpoint will be parasitological response determined as sustained negative qualitative PCR at 24 months after treatment. The proportion of participants with positive qualitative PCR will be measured at 1, 4, 6, 8, 12, 18, and 24 months from end of treatment. The frequency of adverse events leading to treatment discontinuation will be compared. An economic evaluation will be conducted assessing the direct and indirect costs, including procedures associated with the management of adverse events.

ELIGIBILITY:
Inclusion Criteria:o Adults aged ≥ 18 years;

* CD diagnosis through the positivity of two serological tests that use different antigens (recombinant and native antigens, according to World Health Organization (WHO) recommendations) (28).
* Informed consent form read and signed by the participant.
* Weight ≥ 50 kg to ≤ 95 kg.

Exclusion Criteria:

* o Currently pregnant, breastfeeding or expressing gestational desire for the next 2 months.

  * Previously received treatment with Benznidazole (BZN) or NIfurtimox (NFX) - (either completely or incompletely);
  * Any concomitant use or documented history of using allopurinol or antifungals (ketoconazole, itraconazole and posaconazole);
  * History of hypersensitivity, allergic or serious adverse event (SAE) to any "nitroimidazole", and/or its components;
  * Acute or chronic health problems that, in the informed opinion of the investigator, may interfere with the evaluation of the efficacy and/or safety of the drug. Examples are acute infections, Human Immunodeficiency Virus (HIV) infections, liver disease with liver failure and kidney disease requiring support treatment;
  * Signs and/or symptoms of severe cardiac form of CD ;
  * History of cardiomyopathy, heart failure or severe ventricular arrhythmia of any etiology;
  * Alcoholic participants or those with a history of alcohol abuse (considered as intake of >4 drinks on any single day AND >14 drinks per week for men and >3 drinks on any single day AND >7 drinks per week for women);
  * Have basic laboratory parameters outside the normal range or parameters that are considered clinically relevant by the physician responsible for the participant;
  * Participation in another clinical trial over the past 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with sustained negative Polymerase Chain Reaction (PCR) during the 24 months of follow-up after treatment. | during the 24-month follow-up
  The treatment efficacy of each treatment arm is assessed through the proportion of patients with negative parasitaemia measured by PCR during the first 24 months after starting treatment

SECONDARY OUTCOMES:
Incidence of Adverse Events (AE) leading to treatment discontinuation during treatment period | during treatment period (up to 8 weeks)
  The safety profile will me measured with the proportion of patients with treatment discontinuation atributed to the drug toxicity in each treatment arm
Proportion of participants with positive PCR at different time points | At the different time points: 1, 4, 6, 8, 12, 18 and 24 months after the end of treatment
  Parasitic kinetics will be evaluated by detecting parasitic DNA measured by qualitative PCR in peripheral blood in 1, 4, 6, 8, 12, 18 and 24 months after the end of treatment in each of the different therapeutic regimens.

OTHER OUTCOMES:
Incidence and severity of clinically relevant events attributed to Chagas disease | during the 24-month follow-up
  To assess the incidence of events will be taking into account a composite outcome of clinically relevant events: number of hospitalizations, progression to cardiac form or deaths related to Chagas disease.
To measure the quality of life (QoL) of participants | during the 24-month follow-up
  Quality of life will be assessed through longitudinal changes on the score of quality of life using the instrument: The World Health Organization Quality of Life Brief Version (WHOQoL-BREF)
To measure the quality of life (QoL) of participants | during the 24-month follow-up
  Quality of life will be assessed through longitudinal changes on the score of quality of life using the instrument EuroQol 5 Dimensions (EQ5-D)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Israel Molina, Minas Gerais, Belo Horizonte
  - Monique Gurgel de Oliveira, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT06339710/Prot_000.pdf
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT06339710/ICF_001.pdf